CLINICAL TRIAL: NCT05498363
Title: Bacteriophage Therapy of Difficult-to-treat Infections: a Retrospective, Observational Analysis of the First One Hundred Consecutive Cases Facilitated by a Belgian Consortium
Brief Title: Bacteriophage Therapy of Difficult-to-treat Infections
Acronym: BT100
Status: Completed | Type: Observational
Sponsor: Queen Astrid Military Hospital (Other)
Responsible Party: Principal Investigator, Sarah Djebara, Internal Medicine and Infectious Diseases Physician, Queen Astrid Military Hospital
Other Study IDs: BT100
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Bacterial Infections
Keywords: Bacterial infections; Bacteriophages; Antibiotic resistance; Observational study; Retrospective analysis; Difficult to treat infections
MeSH Terms: conditions — Bacterial Infections | interventions — Phage Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Bacteriophage therapy — Difficult-to-treat bacterial infections were treated with bacteriophages (selected from a collection of 25 individual bacteriophages and 6 bacteriophage cocktails), which were shown to target the patient's infecting bacterial strain (in vitro)

SUMMARY:
A retrospective, observational analysis of the first one hundred consecutive cases of bacteriophage therapy of difficult-to-treat infections, facilitated by a Belgian consortium.

DETAILED DESCRIPTION:
Background: In 2008, the Queen Astrid military hospital (QAMH) re-initiated treatments with phages, in selective cases. The QAMH implemented a Phage Therapy Coordination Center (PTCC), which is an essential step in the re-introduction of safe and efficient phage therapy, in collaboration with several hospitals and the public health authorities.

In 2018, Belgium implemented a pragmatic phage therapy framework that centers on the magistral preparation (compounding pharmacies in the US) of tailor-made phage medicines, which paved the way for a broader and more structured application of phages in Belgium.

The PTCC facilitated phage therapy in about 110 difficult-to-treat infections in patients in Belgium, but also abroad, as the Belgian is increasingly finding appeal in other European countries.

Objective: The goal of this study is to retrospectively analyse observational data on the first one hundred consecutive phage therapy cases of difficult-to-treat infections, which were facilitated by the PTCC. The knowledge gained from these cases would help physicians to select effective treatment protocols and to design new clinical trials.

Study design: A de-identified database consisting of demographical, microbiological and clinical observational data on 100 consecutive phage applications performed between 01/01/2008 and 31/05/22 will be retrospectively analyzed. A list of the parameters that will be analyzed can be found in addendum 1.

According to the EU Regulation No 536/2014 (Clinical Trials Regulation) and its transposition to Belgian Law, the retrospective non-interventional study of the de-identified existing phage therapy database is not considered as a an experiment on the human person and does not require informed consent.

The R software environment will be used to analyze the correlation between treatment variables, including the applied phage products (used in combination with antibiotics or not), clinical protocols (proposed by the PTCC, and mostly based on the experiences of the Eliava Institute in the Republic of Georgia), infection types, possible adverse events, clinical outcome (improvement or not), and microbial eradication.

Results will be translated into practical recommendations, which will help physicians to select effective treatment protocols and to design new clinical trials.

The quality control of the used phage products was performed by Sciensano (formerly known as the Belgian Scientific Institute for Public Health) and clinical applications were performed in 34 hospitals in 12 countries (Belgium, United Kingdom, Germany, France, The Netherlands, Switzerland, Latvia, Tunisia, Spain, Portugal, Italy and Austria), under four different regulatory frameworks:

1. Standard of care with magistral phage preparations (since 2018)
2. Article 37 (unproven interventions in clinical practice) of the Declaration of Helsinki
3. Standard of care with unlicensed medicines (in the United Kingdom)
4. "Autorisation Temporaire d'Utilisation" (ATU) (in France) Written informed consent for the clinical application of phages was obtained from the involved patients or their legal representatives according to local provisions. Where warranted, local ethical committee approval for the application of phage therapy was obtained.

The data was obtained through the patients' treating physicians and their authorisation to analyse this data, and a possible scientific publication of the results of this study, will be obtained.

The study is conducted at the QAMH in Brussels under the responsibility and supervision of Dr. Sarah Djebara of the PTCC of the QAMH.

Addendum 1. Observational data on the 100 consecutive phage therapy cases

Demographics*:

Country in which the therapy was performed/ Year in which phage therapy was initiated/ Patient gender/ Patient age

Infection:

Primary infection type/ Secondary infection type/ Acute or chronic infection?/ Additional relevant information/ Organisms/ Antibiotic resistance profile of the targeted strain(s)

Phage product:

Phage name(s)/ Diluent/ Concentration (pfu/ml)

Treatment:

Intraoperative application/ Application route 1 (Dose/Duration)/ Application route 2 (Dose/Duration)/ Concomitant antibiotic treatment/ Ambulatory or hospitalized?

Adverse events:

Adverse event/Duration/Severity/Relationship to phage treatment?/Action

Clinical outcome:

Clinical improvement?/Microbial eradication?/Clinical comment (additional relevant information)

Regulatory context

Published case? If yes, reference

* The demographics data are separated from the individual cases

ELIGIBILITY:
Inclusion Criteria:

* Patients with difficult-to-treat bacterial infections

Exclusion Criteria:

* None

Ages: 1 Month to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with difficult-to-treat bacterial infections for which bacteriophage therapy was requested by the treating physician, and considered to be feasible and potentially beneficial by the Phage Therapy Coordination Center (PTCC) of the Queen Astrid military hospital (QAMH)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | One week to one year after treatment, depending on the infection type
  Clinical improvement of at least one symptom associated with the original bacterial infection, as assessed by the treating physician
Microbial eradication | One week to one year after treatment, depending on the infection type
  The absence of the original causative agent of the bacterial infection in culture
Adverse reactions | One week to one year after treatment, depending on the infection type
  Duration and severity of adverse reactions, as assessed by the treating physician

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Djebara, MD, Principal Investigator — Queen Astrid Military Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pirnay JP, Djebara S, Steurs G, Griselain J, Cochez C, De Soir S, Glonti T, Spiessens A, Vanden Berghe E, Green S, Wagemans J, Lood C, Schrevens E, Chanishvili N, Kutateladze M, de Jode M, Ceyssens PJ, Draye JP, Verbeken G, De Vos D, Rose T, Onsea J, Van Nieuwenhuyse B; Bacteriophage Therapy Providers; Bacteriophage Donors; Soentjens P, Lavigne R, Merabishvili M. Personalized bacteriophage therapy outcomes for 100 consecutive cases: a multicentre, multinational, retrospective observational study. Nat Microbiol. 2024 Jun;9(6):1434-1453. doi: 10.1038/s41564-024-01705-x. Epub 2024 Jun 4. PMID 38834776